CLINICAL TRIAL: NCT04472299
Title: Paravertebral Block to Reduce the Incidence of New Onset Atrial Fibrillation After Cardiac Surgery: A Prospective Randomized Controlled Pilot Trial
Brief Title: Paravertebral Block to Reduce the Incidence of New Onset Atrial Fibrillation After Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANES-2020-28859
Record Dates: First submitted 2020-07-09; First posted 2020-07-15 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: New Onset Atrial Fibrillation; Anesthesia, Local; Cardiac Disease
MeSH Terms: conditions — Heart Diseases | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Participants in this group will receive the intervention.
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution
- Control (No Intervention): Participants in this group will receive no intervention.

INTERVENTIONS:
Drug: Ropivacaine 0.2% Injectable Solution — Patients in the intervention group will have ultrasound guided bilateral T3 paravertebral catheters placed prior to surgery. Prior to surgery, these patients will have 5ml of 1.5% lidocaine with 1:200,000 epinephrine injected in each catheter. Ropivacaine 0.2% will be administered via programmed intermittent bolus of 7ml every 60 minutes through each catheter during and after surgery.
  Arms: Experimental

SUMMARY:
The purpose if this pilot study is to determine if a perioperative infusion of 0.2% ropivacaine via bilateral T3 paravertebral catheters can decrease the incidence of new onset atrial fibrillation following primary CABG and/or valve surgery and compare a number of secondary outcomes.

DETAILED DESCRIPTION:
Patients in the intervention group will have ultrasound guided bilateral T3 paravertebral catheters placed prior to surgery. Prior to surgery, these patients will have 5ml of 1.5% lidocaine with 1:200,000 epinephrine injected in each catheter. Ropivacaine 0.2% will be administered via programmed intermittent bolus of 7ml every 60 minutes through each catheter during and after surgery. Patients in the control group will receive no block and undergo surgery with routine anesthetic care guided by their cardiac anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

- Participants must be undergoing one of the following elective or urgent (but not emergent) surgeries: A) Primary Coronary Artery Bypass Graft (CABG) B) Primary Surgical Aortic Valve Replacement (sAVR) C) Primary Surgical Mitral Valve Replacement (sMVR) D) Combined CABG & surgical valve replacement

Exclusion Criteria:

* History of atrial fibrillation or flutter
* Infective endocarditis
* Left ventricular ejection fraction (LVEF) < 30%
* Emergency surgery
* Redo surgery
* Contraindication to block placement including local anesthetic allergy, bleeding diathesis (physiologic or iatrogenic)
* Body mass index > 35kg/m2
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Incidence of New-Onset Atrial Fibrillation (NOAF) | 5 days
  The primary outcome for this trial is the incidence of new-onset atrial fibrillation (NOAF) in the first 5 days following cardiac surgery, defined as atrial fibrillation and/or flutter as recorded on a 12-lead ECG or rhythm strip for greater than 30 seconds in patients with no prior history of atrial fibrillation and/or flutter. Outcome is reported as the percent of participants with NOAF in each arm.

SECONDARY OUTCOMES:
Cumulative Opioid Use - Average Dosages | 24, 48, 72, 96, and 120 hours post-operatively
  Outcome reported as the average opioid dosage at 24, 48, 72, 96, and 120 hours post-operatively.
Cumulative Opioid Use - Morphine Equivalents | 24, 48, 72, 96, and 120 hours post-operatively
  Outcome reported as the cumulative opioid use in morphine milligram equivalents at 24, 48, 72, 96, and 120 hours post-operatively.
Time to Extubation | approximately 5 days
  Outcome reported as the amount of time (in hours) participants remain intubated post-operatively.
Intensive Care Unit (ICU) Length of Stay | approximately 5 days
  Outcome reported as the length of time (in days) that participants are admitted to the intensive care unit (ICU) post-operatively.
Hospital Length of Stay | approximately 7 days
  Outcome reported as the length of time (in days) that participants remain admitted to the hospital post-operatively.
30-Day Mortality | 30 days
  Outcome reported as the percent of participants in each arm who expire in the 30 days following surgery.
Cumulative ICU sedation doses | 24 and 72 hours post-operatively
  Outcome reported as the cumulative doses of sedatives (Midazolam, Fentanyl, Propofol, Dexmedetomidine, Haloperidol, Olanzapine) at 24 hours and 72 hours post-operatively.
Diagnosis of delirium during index hospitalization | approximately 7 days
  Outcome reported as the percent of participants in each arm who are diagnosed with delirium during hospital admission.
Quality of Recovery 15 (QOR-15) Scores | 24, 48, 72, 96, and 120 hours post-operatively
  The Quality of Recovery 15 is a 15-item survey evaluating recovery after surgery and anaesthesia. Items are rated on a scale 0-10. Total scores are a sum of item scores and range 0-150, with higher scores representing a higher quality of recovery.
Average pain score | 24, 48, 72, 96, and 120 hours post-operatively
  Participants will be asked to rate their pain on a scale from 0 (no pain) to 10 (maximum pain imaginable).
Block-associated complications | approximately 5 days
  Outcome reported as the number of block-associated complications including catheter infection, vascular puncture, bleeding that results in neurologic compromise, pneumothorax.
Block performance time | approximately 1 hour
  Outcome reported as the length of time (in minutes) for placement of catheters.
Duration of vasopressor requirement | approximately 24 hours
  Outcome reported as the length of time (in hours) that participants require vasopressor therapy.

CONTACTS AND LOCATIONS:
Overall Officials: James Flaherty, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No